CLINICAL TRIAL: NCT02026518
Title: Effect of Cholecalciferol, Soy Isoflavones in Patients With Irritable Bowel Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mahsa Jalili, Mrs, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 459
Record Dates: First submitted 2013-12-26; First posted 2014-01-03 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Irritable Bowel Disease
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Soybean Proteins; Cholecalciferol; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Soy (Experimental): Group Soy receiving placebo similar to 50000 IU cholecalciferol (includes MCT oil) biweekly for 6 weeks in addition to 40 milligram (2 capsules per day) soy isoflavones capsules for 6 weeks
  Interventions: Dietary Supplement: Soy isoflavones; Dietary Supplement: placebo of cholecalciferol
- Soy- Cholecalciferol (Experimental): Group Soy- Cholecalciferol receiving Supplement in form of 40 milligrams soy isoflavones (diadzein, genistein, glycitin) per day (2 capsules of 20 milligrams) for 6 weeks in addition to supplement of cholecalciferol (vitamin D3) biweekly for 6 weeks
  Interventions: Dietary Supplement: Soy isoflavones; Dietary Supplement: cholecalciferol
- Placebo (Placebo Comparator): Group Placebo receiving Placebo in similar form of cholecalciferol supplement biweekly for 6 weeks in addition to 40 milligrams placebo in similar form of soy isoflavones including starch for 6 weeks
  Interventions: Dietary Supplement: Placebo of soy isoflavones; Dietary Supplement: placebo of cholecalciferol
- Cholecalciferol (Experimental): Group Cholecalciferol receiving oral Placebo in similar form to soy isoflavones (diadzein, genistein, glycitin) supplement including starch (2 capsules per day) for 6 weeks in addition to 50000 IU cholecalciferol supplement biweekly for 6 weeks
  Interventions: Dietary Supplement: cholecalciferol; Dietary Supplement: Placebo of soy isoflavones

INTERVENTIONS:
Dietary Supplement: Soy isoflavones
  Arms: Soy; Soy- Cholecalciferol
Dietary Supplement: cholecalciferol
  Other Names: Vitamin D
  Arms: Cholecalciferol; Soy- Cholecalciferol
Dietary Supplement: Placebo of soy isoflavones
  Arms: Cholecalciferol; Placebo
Dietary Supplement: placebo of cholecalciferol
  Arms: Placebo; Soy

SUMMARY:
Fasting blood specimens will be taken from the patients with IBS that have inclusion criteria. First, the objectives and method of study will be explained to the patients and informed consent form will be taken from them. They will be divided into 4 groups by an adjusted randomized blocking and the clinical outcomes, quality of life, emotional stress questionnaires will be completed before and after intervention. During 6 weeks, they will receive 2 capsules of soy isoflavones per day, 50000IU vitamin D biweekly in addition to the other placebo form, both of them and placebo of both. At the end, body mass index ( BMI), serum TNF-Alpha, TAC, gene expression of GATA3, ROR gamma, FOXP3 in lymphocytes and gut permeability will be measured. The quantity of polymorphisms of vitamin D and estrogen receptors will be determined.

ELIGIBILITY:
Inclusion Criteria:

1. age 18-75 yrs
2. patients with Irritable Bowel Syndrome (IBS) according to ROME III criteria
3. BMI 18-25
4. a- no intestinal organic diseases b- no intestinal infection c- no history of chronic gastrointestinal and colorectal diseases d- no intestinal major surgery
5. no regular use of antibiotics, anti-constipation and anti-diarrhea, immune suppressors, metoclopramide, cisapride, diphenoxylate, opium and non-steroidal anti-inflammatory drugs
6. no pregnancy and lactation
7. not athlete or bed rest
8. no history of breast cancer in herself or her family
9. no severe psychosis

Exclusion Criteria:

1. a- use of soy isoflavones or vitamin D one year before the study b- use of soy milk or soy nuts during study
2. diet changes during study
3. use of artificial sweetener 2 days before study
4. no desire to complete the study
5. adverse effect of supplement
6. pregnancy during study

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-01; Primary Completion 2014-04 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Clinical Outcomes (pain, flatulence, diarrhea, constipation ) at 6 weeks | 6 weeks

SECONDARY OUTCOMES:
Change of baseline in gut permeability as efficacy at 6 weeks | 6 weeks
Change of baseline in antioxidant status as efficacy at 6 weeks | 6 weeks
Change of baseline in inflammation status as efficacy at 6 weeks | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Gastrointestinal Clinics of Tehran University of Medical Sciences, Tehran, Tehran Province, Iran

REFERENCES:
- [Derived] Jalili M, Vahedi H, Poustchi H, Hekmatdoost A. Soy isoflavones and cholecalciferol reduce inflammation, and gut permeability, without any effect on antioxidant capacity in irritable bowel syndrome: A randomized clinical trial. Clin Nutr ESPEN. 2019 Dec;34:50-54. doi: 10.1016/j.clnesp.2019.09.003. Epub 2019 Oct 2. PMID 31677711
- [Derived] Jalili M, Hekmatdoost A, Vahedi H, Poustchi H, Khademi B, Saadi M, Zemestani M, Janani L. Co-Administration of Soy Isoflavones and Vitamin D in Management of Irritable Bowel Disease. PLoS One. 2016 Aug 4;11(8):e0158545. doi: 10.1371/journal.pone.0158545. eCollection 2016. PMID 27490103
- [Derived] Jalili M, Vahedi H, Janani L, Poustchi H, Malekzadeh R, Hekmatdoost A. Soy Isoflavones Supplementation for Patients with Irritable Bowel Syndrome: A Randomized Double Blind Clinical Trial. Middle East J Dig Dis. 2015 Jul;7:170-6. PMID 26396720